CLINICAL TRIAL: NCT06722742
Title: Frequency of Shivering Among Patient Treaed With IV Tramadol Versus Iv Ketamine in Prevention of Post Spinal Anesthesia Undergoing Cesarean Section: Rendomiced Control Trial
Brief Title: Use of Iv Tramadol and Ketamine for Prevention of Post Spinal Anesthesia Shivering
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Liaquat National Hospital & Medical College (Other)
Responsible Party: Principal Investigator, Nazish Kanwal, Principal Investigator, Liaquat National Hospital & Medical College
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: #882-2023-LNH-ERC
Record Dates: First submitted 2024-11-28; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Shivering, Spinal Anesthesia
Keywords: shivering; Spinal anesthesia; Ketamine; Tramadol and Metclopromide
MeSH Terms: interventions — Tramadol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group K (Active Comparator): Group K receive Inj: ketamine
  Interventions: Drug: Ketamine only
- Group T (Active Comparator): Group T receive Inj: Tramadol
  Interventions: Drug: Tramadol

INTERVENTIONS:
Drug: Ketamine only — Inj: Ketamine given to group K following spinal anesthesia
  Arms: Group K
Drug: Tramadol — Inj Tramadol given to group T following spinal anesthesia
  Arms: Group T

SUMMARY:
*Ketamine:* Ketamine is a medication that can help reduce shivering by blocking certain nerve signals in the brain. It's like a "nerve blocker" that helps calm down the body's shivering response.

- *Tramadol:* Tramadol is a pain medication that can also help reduce shivering. It works by affecting the brain's temperature regulation centers, which helps to reduce the shivering response.

DETAILED DESCRIPTION:
Post-spinal shivering is when a patient starts shaking or shivering after receiving spinal anesthesia. This can be uncomfortable and even scary for the patient.

Using ketamine and tramadol to reduce post-spinal shivering can have several benefits, including:

* Reduced discomfort and anxiety for the patient
* Improved patient satisfaction
* Reduced need for additional medications or interventions
* Faster recovery times

ELIGIBILITY:
Inclusion Criteria:

* Pateint for elective cesarean section
* Age 18 to 40 years
* ASA 1 and 2

Exclusion Criteria:

* ASA 2 and 3
* Cesarean section requiring general anesthesia
* Hypersensitivity to Ketamine, Tramadol and Opiods
* History of cardiovascular disease

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Shivering | 20 minutes to 12 hours
  Scale validated by crossley and mahajan Grade 0: No shivering Grade 1: Piloerection, peripheral vasoconstriction, peripheral cyanosis, or mild fasciculation of the face or neck, but no visible muscle activity Grade 2: Visible muscle activity in one muscle group Grade 3: Visible muscle activity in more than one muscle group Grade 4: Gross muscle activity involving the entire body

CONTACTS AND LOCATIONS:
Overall Officials: Nazish Dr Nazish Kanwal, Principal Investigator — Liaquat national hospital and medical college
Locations (1):
- Liaquat National Hospital and Medical College, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
Patient confidentiality*: Sharing IPD could compromise patient confidentiality and anonymity, potentially harming participants or their families.
  * Informed consent*: Participants may not have provided informed consent for their data to be shared, which could raise ethical concerns.

REFERENCES:
- See also: The effect of ketamine versus tramadol on prophylactic post-spinal shivering in those patients undergoing orthopedic surgery: a prospective cohort study design, 2020 Ashebir Debalike Gemechu 1, Tsegaye Demeke Gebremedhin 1,✉, Andualem Assefa Andebiku 1, — https://pmc.ncbi.nlm.nih.gov/articles/PMC9685948/